CLINICAL TRIAL: NCT02872415
Title: Impact of Alternative Blood Glucose Testing Site (Forearm) on Pain Reduction in Preterm Neonates.
Brief Title: Effect of Site on Pain in Preterm Neonates
Acronym: NOBOBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2016-18; 2016-A01349-42 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Great Premature Newborn

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The forearm as blood puncture site (Experimental): The child receives a puncture blood on the forearm
  Interventions: Biological: Blood puncture site
- Fingers like blood puncture site (Placebo Comparator): Premature receiving a puncture blood on the finger
  Interventions: Biological: Blood puncture site

INTERVENTIONS:
Biological: Blood puncture site — Blood puncture site

SUMMARY:
Numerous experimental and clinical studies have shown that preterm neonates are particularly sensitive to stress. Preterm neonates routinely undergo painful invasive procedures. Each situation causing pain or discomfort can alter their development and cause short term cardiovascular consequences but also have long-term neurocognitive influences. Repetitive procedural pain can also lead to changes in the pain sensitivity threshold therefore. The most common painful procedures are lancing for blood glucose testing. In adults, infants and term newborns, forearm blood glucose testing has been demonstrated to be less painful than conventional sites (heel, fingers). But data is lacking in preterm neonates.

The primary purpose of this study is to demonstrate a significant reduction in pain response during forearm blood lancing vs conventional sites (fingers, heel) in preterm neonates born up to 32 weeks gestation.

This study is an interventional multicenter (3 centers), randomized, double bind trial with a cross over assignment. 60 premature neonates born between 23 to 32 weeks.

Gestation with a postnatal age less than 72 hours that will undergo at least 3 blood glucose pricks will be included. The different sites will be randomly successively tested.

ELIGIBILITY:
Inclusion Criteria:

* Premature neonates 23 to 32 weeks gestation
* Infant born with a postnatal age greater than or equal to 3 hours and less or equal to 72 hours
* Infant born with at least 3 blood glucose testing in less than 72 hours

Exclusion Criteria:

* Severe congenital anomalies that could alter pain perception or expression
* Extremities congenital anomaly impeding blood glucose testing on different sites
* Infants born to mothers known to be receiving opiates
* Severe haemodynamic disturb
* Severe neurologic injury
* Neonate with opioids or sedatives medications
* No parental consent

Ages: 3 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
The pain assessment | 12 months
  Painful response using Premature Infant Pain Profile (PIPP)

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No